CLINICAL TRIAL: NCT06718881
Title: Investigation of the Effect of Virtual Reality Environment on Developing Clinical Skills in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gülçin NACAR, Associate professor, Inonu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: TUBİTAK 1001
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: University Students
Keywords: Nursing; Virtual Reality Environment; Case Discussion; Role Playing; The Presence Questionnaire; Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental model
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the project, theoretical lessons were given on preeclampsia, postpartum care, and condom counseling, each in a separate week. After each theoretical lesson, an application was made in the laboratory on the subject explained in the same week. The applications were made in the form of a simulation application in a virtual reality environment for the students in the experimental group.
  Interventions: Other: simulation application in a virtual reality environment
- Control (No Intervention): After classical training, case discussion and role play were conducted.

INTERVENTIONS:
Other: simulation application in a virtual reality environment — In the project, theoretical lessons were given on preeclampsia, postpartum care, and condom counseling, each in a separate week. After each theoretical lesson, an application was made in the laboratory on the subject explained in the same week. The applications were made in the form of a simulation application in a virtual reality environment for the students in the experimental group.
  Arms: Intervention

SUMMARY:
To reduce the negative consequences of these problems in clinical practice on the quality of education in the nursing profession, laboratory applications of vocational courses in undergraduate education have become more important. In this context, the research aimed to determine the use of a virtual reality application, an innovative training method to increase the quality of nurses' clinical practice training, in the Obstetrics-Gynecology and Diseases Nursing (DKSH) course and its effect on students' course success. I

DETAILED DESCRIPTION:
When considering the duties and responsibilities of nurses in the health system, it is necessary to train well-educated, professional nurses to ensure patient safety and quality of care. However, nurses' many problems with their clinical practice are important obstacles to getting a good education. To reduce the negative consequences of these problems in clinical practice on the quality of education in the nursing profession, laboratory applications of vocational courses in undergraduate education have become more important. In this context, the research aimed to determine the use of a virtual reality application, an innovative training method to increase the quality of nurses' clinical practice training, in the Obstetrics-Gynecology and Diseases Nursing (DKSH) course and its effect on students' course success. In the study, the virtual reality application was prepared for preeclampsia, postpartum care and condom counseling, which are the most frequently encountered by students in professional practice and are of great medical importance. In addition, the effect of simulation training in the virtual reality environment on the student's decision-making self-confidence and anxiety in real clinical practice was also evaluated. In this context, the research aims to determine the effect of a virtual reality environment on improving clinical skills in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older, taking the Obstetrics, Gynecology and Obstetrics Nursing course for the first time, attending the course and taking the information technology course.

Exclusion Criteria:

* Being visually or hearing impaired, graduating from a health vocational high school, arriving late or leaving early for case discussions or role-play scenarios, and staying in the virtual environment for less than 5 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Self-confidence in Clinical Decision Making in Nursing | 3 month
  The median score of self-confidence in Clinical Decision Making in Nursing was 127.00 (CAG: 30.00) in the experimental group and 112.00 (CAG: 36.00) in the control group (p<0.05).
Anxiety in Clinical Decision Making in Nursing | 3 month
  The mean score of anxiety in Clinical Decision Making in Nursing was 52.00 (CAG: 24.00) in the experimental group and 60.00 (CAG: 35.00) in the control group (p<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Nacar, PHD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Battalgazi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' data were collected for research purposes only according to the ethical principle of confidentiality and protection. Therefore, it cannot be shared.